CLINICAL TRIAL: NCT00582127
Title: Evaluation of a Handheld Evoked Response Potentials (ERP) System as an Effective Method to Diagnose Alzheimer's Disease
Brief Title: Evaluation of the COGNISION(TM) System as an Event-related Potential (ERP) Collection System.
Status: Completed | Type: Observational
Sponsor: Neuronetrix, Inc. (Industry)
Collaborators: University of Kentucky (Other)
Responsible Party: Charles D. Smith, M.D., University of Kentucky
Other Study IDs: VAL-UK-01
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Alzheimer's Disease
Keywords: senile; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Mild-moderate Alzheimer's Disease
- 2: Age-matched Controls

SUMMARY:
This study will evaluate a handheld event-related potential (ERP) testing device from Neuronetrix, Inc. as a method to collect ERP data in an outpatient setting.

An ERP system records electrical signals at the scalp that are produced by the brain when performing cognitive tasks. By doing this study, we hope to evaluate various performance parameters of the COGNISION(TM) system.

DETAILED DESCRIPTION:
Patients who have a current diagnosis of mild-moderate dementia and suspected of having Alzheimer's disease (AD) along with cognitively normal age-matched controls will be recruited for this study. The Alzheimer's subjects either will have had a complete clinical and neuropsychiatric workup or will have those tests performed during the study.

Both groups, AD and controls will be asked to listen to a series of sounds and press a button on a handheld control box when a target sound is heard. The COGNISION(TM) headset on each subject's head will then record the electrical signals during this task.

Four important features of the COGNISION(TM) will be investigated:

1. Patient tolerance
2. Ease of use
3. Data quality
4. Network architecture

ELIGIBILITY:
Inclusion Criteria for AD:

* Age 60 to 85
* Mild to moderate diagnosis of Alzhiemer's disease

Inclusion Criteria for Control:

* Age 60 to 85
* Cognitively healthy with no complaints

Exclusion Criteria:

* Subjects with advanced AD and severe impairment (CDR > 2, MMSE less than 15)
* Neurological disorders such as stroke, Parkinson's disease, Huntington's disease, multiple sclerosis, brain tumor, delirium, or psychiatric disorder other than depression (e.g. schizophrenia)
* Subjects with life threatening illnesses and subjects with significant hearing or visual impairments
* Subjects with a current prescription for psychoactive pharmaceuticals

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and family from the University of Kentucky Sanders Brown Center for Aging
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Signal to noise ratio (SNR) of ERPs | 9 months

SECONDARY OUTCOMES:
Patient tolerance of the COGNISION(TM) system. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Smith, M.D., Principal Investigator — University of Kentucky
Locations (1):
- Sanders Brown Center for Aging, Neurology Dept., Lexington, Kentucky, United States

REFERENCES:
- [Background] Polikar R, Topalis A, Green D, Kounios J, Clark CM. Comparative multiresolution wavelet analysis of ERP spectral bands using an ensemble of classifiers approach for early diagnosis of Alzheimer's disease. Comput Biol Med. 2007 Apr;37(4):542-58. doi: 10.1016/j.compbiomed.2006.08.012. Epub 2006 Sep 20. PMID 16989799
- See also: Website for manufacturer of COGNISION(tm) System being tested — http://www.neuronetrix.com